CLINICAL TRIAL: NCT03726840
Title: Sensory-based Stimulation to Increase Alertness and Behavioral Performance During Simulated Driving
Brief Title: Sensory Stimulation During Simulated Driving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2018-2204
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Behavior
MeSH Terms: conditions — Behavior | interventions — Odorants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Driving performance no fragrance (No Intervention): healthy young (ages 24-35 years) and older (ages 60-85 years) with no fragrance
- Driving performance Fragrance (Experimental): healthy young (ages 24-35 years) and older (ages 60-85 years) with fragrance
  Interventions: Other: Fragrance

INTERVENTIONS:
Other: Fragrance — peppermint, rosemary, and zest/pulp will increase memory recall for navigation and improve reaction times for braking, compared to performance during unscented conditions
  Arms: Driving performance Fragrance

SUMMARY:
The purpose of this study is to examine the effect of three specific odors on simulated driving performance. It is hypothesized that the presence of peppermint, rosemary, and zest/pulp will increase memory recall for navigation and improve reaction times for braking, compared to performance during unscented conditions

DETAILED DESCRIPTION:
This study will examine the effect of scented odors on the attention and behavioral performance of healthy young adult and older adult drivers. Past research indicates that specific scented odors (i.e., peppermint and cinnamon) enhance motivation, performance and alertness, decrease fatigue and stimulate the central nervous system in a variety of contexts. The current study will examine the effect of three different odors on simulated driving as participants perform navigation and braking scenarios. This study will be the first of its kind to elucidate the association between specific scents and performance gains in simulated driving. The data will serve as proof-of-concept for eventual patient focused interventions relative to sensory stimulation and driving.

ELIGIBILITY:
Inclusion Criteria:

* valid drivers license
* normal or corrected to normal vision

Exclusion Criteria:

* no drivers license
* hyperopic vision without contact lenses
* history of congenital or acquired cognitive, ophthalmologic, or neurological disorders including developmental delay, brain tumor, stroke, or known peripheral or central vestibular disorders
* participants who have been diagnosed with Attention Deficit Hyperactivity Disorder (ADHD) will be excluded
* Participants will also be excluded if they have: (a) a history of skin irritation or sensitivity to scented products or cosmetics, (b) known skin allergies, sensitive skin or allergies to fragrance, (c) suffers from a cold, allergy, sinus condition or any other condition that might interfere with their sense of smell and (d) is pregnant or nursing.
* Participants will also be excluded if they smoke or use tobacco related products
* participants will be excluded if they commonly experience motion sickness

Ages: 24 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Navigation Assessment | 30 minutes
  The navigation task will consist of up to six blocks of instruction/recall segments that will contain the same number of turns over the same distance, but with novel environmental stimuli and a randomized order of turns unique to each block.

SECONDARY OUTCOMES:
Braking Assessment | 15 minutes
  a virtual stop sign will appear suddenly in the middle of the visual field. The participant will be instructed to come to a stop as quickly as possible and to remain stopped until the stop sign disappears
Workload and mood assessment | 5 minutes
  participants will be asked to rank their perceived mental, physical, and temporal demands in combination with their performance, effort and frustration
Scent assessment | 5 minutes
  A short fragrance questionnaire will be given after each study session, in order to ensure that participants are able to distinguish between non-scented and scented conditions

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinanti Childrens Hospital Medical Center, Cincinnati, Ohio, United States